CLINICAL TRIAL: NCT01585532
Title: Evaluation of Various Methods for the Detection of Mycobacterium Tuberculosis Nucleic Acid
Brief Title: Alere Mycobacterium Tuberculosis Urine Study
Status: Completed | Type: Observational
Sponsor: Research Center Borstel (Other)
Collaborators: Alere Technologies GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: RCBorstel002; CLDG-0402 (Other: Alere Technologies GmbH)
Record Dates: First submitted 2012-04-13; First posted 2012-04-26 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Urine; Nucleic acid; Alere; Borstel
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Sputum Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TB suspects with alternative final diagnosis
- Confirmed tuberculosis patients

SUMMARY:
Current molecular methods will be evaluated for the detection of Mycobacterium tuberculosis specific nucleic acid in urine and blood of patients.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed tuberculosis
* Age >18 years
* informed consent obtained

Exclusion Criteria:

* Previous participation in the study
* Simultaneous participation in a clinical trial investigating a new drug
* Inability to give consent
* Member of a vulnerable study population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or confirmed tuberculosis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity | On admission to hospital
  ROC analysis to determine the best specificity and sensitivity to differentiate between patients with tuberculosis and patients with an alternative diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center Borstel, Borstel, Schleswig-Holstein, Germany